CLINICAL TRIAL: NCT01167140
Title: Cryo-Touch II for the Treatment of Wrinkles
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS-4000
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Results first posted 2012-10-01 (Estimated); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Facial Wrinkles

ARMS (1):
- Cryo-Touch II (Experimental)
  Interventions: Device: Cryo-Touch II

INTERVENTIONS:
Device: Cryo-Touch II — Percutaneous treatment with the device

SUMMARY:
This is a prospective, non-randomized study to evaluate the performance of the MyoScience Cryo-Touch II device for the treatment of wrinkles.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-70 years
* Subject has a glabellar and/or forehead wrinkle rating by investigator of at least 1 at rest on the 5-point Wrinkle Scale (5WS)*
* Subject has signed IRB-approved informed consent form

Exclusion Criteria:

* Subject takes any medication or dietary supplement regularly that affects blood clotting (e.g., Coumadin, aspirin, clopidogrel) or increases the risk of bleeding/bruising
* Subject has had prior surgery that alters the subcutaneous anatomy of the target treatment sites
* The investigator is unable to substantially lessen facial lines by physical separation
* Subject has undergone another facial cosmetic procedures at or above the level of the cheekbones within the past 6 months
* Subject is participating in another facial cosmetic research study

Patient has any of following conditions:

* History of facial nerve palsy
* Marked facial asymmetry
* Ptosis
* Excessive dermatochalasis
* Deep dermal scarring
* Thick sebaceous skin
* History of neuromuscular disorder
* Chronic dry eye symptoms
* Allergy or intolerance to lidocaine

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Aesthetics Research Center, Redwood City, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group
Started | 42
Completed | 41
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Effectiveness and Safety Success
Description: * Effectiveness success: an improvement in line severity in the target area in animation at 30 days post-treatment as rated by the investigator using the 5-point wrinkle scale
  * Safety success: the absence of a device-related serious adverse event (DSAE)
Time Frame: Up to 4 months
Population: All subjects treated were analyzed to the safety endpoint.
Measure: Number; unit: participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 41
participants
  Effectiveness Success (n=36) | 30
  Safety Success (n=41) | 41

2. Secondary Outcome: Participants With One Point Improvement in Line Severity
Description: • Investigators' rating of line severity improvement in the target area in animation at 7 days post-treatment, and at 30-day intervals for 120 days after treatment from baseline
Time Frame: Baseline and up to 4 months
Population: Of the 41 subjects treated, 5 were treated at a lower dose and excluded from the effectiveness measure.
Measure: Number; unit: participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 36
participants
  7 days post-treatment | 32
  60 days post-treatment | 19
  90 days post-treatment | 9
  120 days post-treatment | 2

3. Secondary Outcome: Participants With an Improvement in Global Appearance
Description: • Subjects' global assessment of change in appearance of target area at 7 days post-treatment, and at 30-day intervals for 120 days after treatment to baseline
Time Frame: Up to 4 months
Population: 5 subjects were excluded from effectiveness analysis because they received a lower dose.
Measure: Number; unit: participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 36
participants
  7 days post-treatment | 34
  30 days post-treatment | 32
  60 days post-treatment | 25
  90 days post-treatment | 12
  120 days post-treatment | 2

ADVERSE EVENTS:
Arm/Group | Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 13/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=41)
headache (Nervous system disorders) | 4 (4)
local side effect (Skin and subcutaneous tissue disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other